CLINICAL TRIAL: NCT02939651
Title: A Phase 2, Open-label Study of Pembrolizumab Monotherapy in Patients With Metastatic High Grade Neuroendocrine Tumors
Brief Title: A Study of Pembrolizumab in Patients With Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI-087
Record Dates: First submitted 2016-10-03; First posted 2016-10-20 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Neuroendocrine Tumors
Keywords: Metastatic; High grade
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (Experimental): Monotherapy with PD-1 antibody pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab given intravenously at a fixed dose of 200mg every 3 weeks
  Other Names: Keytruda; MK-3475

SUMMARY:
The purpose of this research study is to test if pembrolizumab is safe and effective for treating patients with metastatic high-grade neuroendocrine tumors who have failed platinum based chemotherapy.The study drug, pembrolizumab has been FDA approved for treating a type of skin cancer called melanoma and for metastatic non-small cell lung cancer. However, it is not approved for treatment of metastatic high-grade neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed metastatic, high grade NET (Ki67 >20%), excluding any high grade NETs of large or small cell type of lung/thymus origin and merkel cell carcinoma
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v. 1.1 as described in detail in section 12.0
3. Has received prior therapy with at least 1 platinum-containing regimen
4. Age > 18 years.
5. ECOG performance status 0 or 1
6. Patients must have normal organ and marrow function
7. Female participants of childbearing potential must have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication). They should also be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
8. Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
9. Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

1. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
3. Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Prior anti-cancer therapy with a monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or not recovered from adverse events (improved to grade 1 or less) due to mAbs administered more than 4 weeks earlier.
5. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks (12 weeks for measurable sites of CNS disease) prior to study Day 1 or not recovered from adverse events (improved to grade 1 or less) due to a previously administered agent. Note: Subjects with neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Known additional malignancy that is progressing or requires active treatment except superficial malignancies of the skin and in situ cervical cancer
7. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
8. Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active non-infectious pneumonitis.
9. Active infection requiring systemic therapy at enrollment.
10. Has a known history of active TB (Bacillus Tuberculosis)
11. Hypersensitivity to pembrolizumab or any of its excipients
12. Has received a live virus vaccine within 30 days of planned start of trial treatment.
13. Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening period through 120 days after the last dose of trial treatment
14. Prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed cell death 1 ligand (PDL-1), anti-PD-L2, or with an agent directed to another co-inhibitory T-cell receptor (e.g. CTLA-4, OX-40, CD137)
15. Known history of human immunodeficiency virus (HIV)
16. Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative]).
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Namrata Vijayvergia, MD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Vijayvergia N, Dasari A, Deng M, Litwin S, Al-Toubah T, Alpaugh RK, Dotan E, Hall MJ, Ross NM, Runyen MM, Denlinger CS, Halperin DM, Cohen SJ, Engstrom PF, Strosberg JR. Pembrolizumab monotherapy in patients with previously treated metastatic high-grade neuroendocrine neoplasms: joint analysis of two prospective, non-randomised trials. Br J Cancer. 2020 Apr;122(9):1309-1314. doi: 10.1038/s41416-020-0775-0. Epub 2020 Mar 10. PMID 32152503

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 56 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: To estimate objective response rate (ORR), using RECIST 1.1, in previously treated metastatic High Grade Neuroendocrine Tumors (HGNET) patients treated with pembrolizumab monotherapy. The Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria will be used for objective tumor response assessment: Complete Response (CR):Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: Upto 3 years
Population: Analysis was completed using data from an external site which accrued 8 patients
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 21
Participants | 1

2. Secondary Outcome: Progression Free Survival (PFS)
Description: To evaluate progression free survival (PFS) (using RECIST 1.1) in metastatic HGNET patients treated with pembrolizumab monotherapy. PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase (at least 5 mm absolute increase) in the sum of the longest diameter of target lesions. PFS was estimated according to the Kaplan-Meier method.
Time Frame: Upto 3 years
Population: Analysis was completed using data from an external site which accrued 8 patients
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 21
weeks | 8.86 [6.00 to 9.43]

3. Secondary Outcome: Overall Survival
Description: To evaluate overall survival (OS) in metastatic HGNET patients treated with pembrolizumab monotherapy. OS was estimated according to the Kaplan-Meier method.
Time Frame: Upto 3 years
Population: Analysis was completed using data from an external site which accrued 8 patients. 95% confidence interval upper limit not estimated
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 21
weeks | 20.43 [12.86 to NA] — Upper band of median survival cannot be estimated

4. Secondary Outcome: Frequency With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Description: Occurence of toxicity, graded according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0.
Time Frame: Upto 3 years
Population: Analysis was completed using data from an external site which accrued 8 patients
Measure: Number; unit: adverse events
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 21
adverse events | 34

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 15/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=21)
Acute kidney injury (Renal and urinary disorders) | 1
Cholangitis (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Polymyaglia (Musculoskeletal and connective tissue disorders) | 1
Elevated ALT (Investigations) | 1
Elevated ALK (Investigations) | 1
Upper GI bleed (Gastrointestinal disorders) | 1
Anemia (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=21)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 3
Anorexia (Psychiatric disorders) | 3
Aspartate aminotransferase increased (Hepatobiliary disorders) | 3
Bloating (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth (General disorders) | 1
Edema limbs (Blood and lymphatic system disorders) | 2
Fatigue (General disorders) | 7
Gastrointestinal disorders (Gastrointestinal disorders) | 1
General disorders and administration site conditions (General disorders) | 2
Hypercalcemia (Endocrine disorders) | 1
Hyperkalemia (Endocrine disorders) | 1
Nausea (General disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rectal pain (Gastrointestinal disorders) | 1
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1
Vomiting (General disorders) | 1

LIMITATIONS AND CAVEATS:
Pembrolizumab can be safely administered to patients with G3NENs but has limited activity as a single agent. Further research to identify active combination therapies should be considered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT02939651/Prot_SAP_000.pdf